CLINICAL TRIAL: NCT04001608
Title: A Phase 3, Multicenter, Open-Label, Single-Arm Study to Investigate the Efficacy and Safety of a 12-Week Regimen of Seraprevir in Combination With Sofosbuvir in Patients With Chronic Genotype 1 Hepatitis C Virus Infection.
Brief Title: Study of Seraprevir in Combination With Sofosbuvir in Chronic Genotype 1 Hepatitis C Virus Infection Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ginkgopharma CO., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GP205-1801
Record Dates: First submitted 2019-06-21; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Seraprevir and sofosbuvir (Experimental): Subjects will receive oral tablets of Seraprevir 100mg twice a day along with oral tablet of sofosbuvir 400 mg,once a day from Day 1 up to Week 12.
  Interventions: Drug: Seraprevir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Seraprevir — Subjects will receive oral tablets of Seraprevir 100 mg, twice a day from Day 1 up to Week 12
  Other Names: GP205
Drug: Sofosbuvir — Subjects will receive oral tablet of sofosbuvir 400 mg, once a day from Day 1 up to Week 12
  Other Names: sovaldi

SUMMARY:
This study was to assess the safety and efficacy of Seraprevir in combination with sofosbuvir administered for 12 weeks in patients with Hepatitis C (HCV) genotype1. Efficacy was assessed by the rate of sustained viral response (SVR) 12 weeks after the discontinuation of therapy (SVR12).

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C virus (HCV) genotype 1 infection (confirmed at screening).
* HCVRNA greater than 10,000 IU/mL at screening.
* Participant must be willing and able to comply with the protocol requirements.
* weight was more than 40 kg.
* age is between 18-75,either sex.

Exclusion Criteria:

* Co-infection with hepatitis B virus or human immunodeficiency virus (HIV).
* Infection with HCV non-genotype 1,or Infection with mixed genotype,or Genotype cannot be confirmed.
* Medical history of major functional organ transplantation.
* Suffering from serious blood system disease(such us Thalassemia/Sickle Cell Anemia).
* Participation in a clinical study within 3 months prior to first dose

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Sustained Virologic Response 12 Weeks After the Actual End of Treatment（SVR12） | Posttreatment Week 12
  SVR12 is defined as HCV RNA < the lower limit of quantification (LLOQ; ie, < 15 IU/mL) 12 weeks following the last dose of study drug.

SECONDARY OUTCOMES:
Percentage of Participants Achieving a Sustained Virologic Response 4 Weeks After the Actual End of Treatment (SVR4) | Posttreatment Week 4
  SVR4 is defined as HCV RNA < LLOQ at 4 weeks following the last dose of study drug.
Percentage of Participants Achieving a On-treatment Virologic Response | week 1,week 2,week 4,week8,week 12
  Percentage of participants who achieved HCV RNA <LLOQ at week 1,week 2,week 4,week8,week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Xuegang Wu, Study Director — Ginkgo Pharma Co., Ltd.
Locations (22):
- China (22):
  - Beijing Ditan Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing YouAn Hospital ,Capital Medical University, Beijing, Beijing Municipality
  - Chongqing Public Health Medical Center, Chongqing, Chongqing Municipality
  - Chongqing Sanxia Center Hospital, Chongqing, Chongqing Municipality
  - Liuzhou General Hospital, Liuchow, Guangxi
  - Affiliated Hospital Of Zunyi Medical University, Zunyi, Guizhou
  - The First Hospital Of Hebei Medical University, Shijiazhuang, Hebei
  - The Sixth People's Hospital Of Zhengzhou, Zhengzhou, Henan
  - Tongji Hospital Affiliated To Tongji Medical College Huazhong University Of Science And technology, Wuhan, Hubei
  - Wuhan Medical Treatment Center, Wuhan, Hubei
  - Wuxi No.5 People's Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital OF Xuzhou Medical University, Xuzhou, Jiangsu
  - The first hospital of JILIN university., Changchun, Jilin
  - The First Affiliated Hospital Of Guangxi Medical University, Guangxi, Nanning
  - First Hospital Of Shanxi Medical University, Taiyuan, Shanxi
  - Traditional Chinese Medical Hospital Affiliated To Southwest Medical University, Luzhou, Sichaun
  - Chengdu Public Health Medical Center, Chengdu, Sichuan
  - Sichuan Province General Hospital, Chengdu, Sichuan
  - First Affiliated Hospital Of Xinjiang Medical University, Ürümqi, Xinjiang
  - Traditional Chinese Medical Hospital Uygur Autonomous Region, Ürümqi, Xinjiang
  - Huzhou Center Hospital, Huzhou, Zhejiang